CLINICAL TRIAL: NCT01161901
Title: Impact of Inflammation Biomarkers on the Acute Respiratory Distress Syndrome Definition in Intensive Care Unit
Brief Title: Impact of Inflammation Biomarkers on the Acute Respiratory Distress Syndrome (ARDS) Definition
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0078
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Plasmatic biomarkers; Lung Morphology; Mechanical ventilation; CT scan
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- blood sample
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — This study's hypothesis is that patients with ARDS criteria and lobar morphology on CT scan present loss of aeration but no inflammatory pulmonary oedema, whereas patients with non lobar morphology on CT scan present both characteristics.
  The primary purpose of our protocol is to show that the patients who respond to ARDS criteria and have a lobar morphology on CT scan do not have an elevation of the biomarkers specific to the pulmonary aggression of ARDS.

SUMMARY:
The ARDS has a clinical definition with criteria of the American-European Consensus Conference (1994). This definition inconveniently applies to a lot of patients with acute respiratory failure.

We know that there are 2 forms of ARDS morphology on CT scan : "lobar attenuation" (loss of aeration with no concomitant excess in lung tissue) predominating in the lower lobes and "non lobar attenuation" with diffuse and massive loss of aeration with excess lung tissue in all the pulmonary parenchyma.

Today, plasmatic biomarkers are used as prognostic and diagnostic markers of ARDS. Some of them are characteristics of the different damages in the ARDS (alveolar epithelium and vascular endothelium lesions) : sRAGE, SP-D, PAI 1 and sICAM 1.

This study's hypothesis is that patients with ARDS criteria and lobar morphology on CT scan present loss of aeration but no inflammatory pulmonary oedema, whereas patients with non lobar morphology on CT scan present both characteristics.

The primary purpose of our protocol is to show that the patients who respond to ARDS criteria and have a lobar morphology on CT scan do not have an elevation of the biomarkers specific to the pulmonary aggression of ARDS.

DETAILED DESCRIPTION:
This multicentric prospective observational study will compare the level of different biomarkers specific to ARDS damages : the soluble form of the receptor for advanced glycation end products (sRAGE), the surfactant protein D (SP-D), Plasminogen Activator Inhibitor type 1 (PAI-1) and Soluble Intercellular Adhesion Molecule-1 (sICAM 1) in the two pulmonary morphologies of ARDS on CT scan : lobar and non lobar.

Patients under mechanical ventilation and with ARDS criteria for less than 24 hours(American-European Consensus Conference, 1994) will be enrolled.

Within 24 hours of enrolment, 10ml of blood sample will be collected and stored at -80°C. Plasmatic biomarker concentrations will be determined through ELISA method.

Within 48 hours of enrolment, patients will have a pulmonary CT scan without injection (end of expiration and ZEEP), a classical practice in this pathology.

Nine university hospitals will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients within the first 24 hours after onset of ARDS according to the 1994 American-European Consensus Conference (AECC)
* Patients under mechanical ventilation

Exclusion Criteria:

* Pregnancy
* Acute exacerbation of diabetes
* Dialysis for end-stage kidney disease
* Alzheimer's disease
* Amyloidosis
* Evolutive neoplastic lesion
* Chronic hepatic disease: type C hepatitis, non alcoholic cirrhosis and adenocarcinoma.
* Evolutive COPD
* Patients enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Defined population
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Plasmatic concentrations of biomarkers specific to the pulmonary aggression of ARDS in the 2 different morphologies on CT scan (lobar and non lobar): • sRAGE • SP-D • sICAM 1 • PAI 1. | within 24 hours of enrolment

SECONDARY OUTCOMES:
Compare the 2 different forms of CT scan morphology in term of : • Mechanical ventilation duration • Mortality at 28 days • Mortality at 90 days | within 48 hours of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France